CLINICAL TRIAL: NCT02912312
Title: Shortening Adjuvant Photon Irradiation to Reduce Edema (SAPHIRE): A Randomized Trial of Hypofractionated Versus Conventionally Fractionated Regional Nodal Irradiation for Invasive Breast Cancer
Brief Title: Hypofractionated vs. Conventional Regional Nodal Radiation Therapy for Patients With Invasive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0142; NCI-2016-01941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0142 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Invasive Breast Carcinoma; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
Keywords: Breast cancer; hypofractionation; radiation therapy; regional nodal irradiation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I: Hypofractionated Regional Nodal Irradiation (RNI) (Experimental): Patients undergo hypofractionated RNI in 15 fractions 5 consecutive days a week for 3 weeks. Patients also undergo additional boost dose of radiation therapy in 5 or 7 fractions on consecutive days following completion of RNI.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II: Standard Regional Nodal Irradiation (RNI) (Active Comparator): Patients undergo standard RNI in 25 fractions 5 consecutive days a week for 5 weeks. Patients also undergo additional boost dose of radiation therapy in 5 or 7 fractions on consecutive days following completion of RNI.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated RNI
  Other Names: Hypofractionated Radiotherapy; hypofractionation
  Arms: Arm I: Hypofractionated Regional Nodal Irradiation (RNI)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo standard RNI
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
  Arms: Arm II: Standard Regional Nodal Irradiation (RNI)

SUMMARY:
To compare how often cancer recurs (comes back) after 3 weeks of radiation compared to 5 weeks of radiation in patients who receive radiation therapy delivered to the lymph nodes near the breast. The side effects that can develop during or after radiation treatment, including how often arm swelling (edema) happens, will also be studied.

DETAILED DESCRIPTION:
Primary Objective: To compare the risk of locoregional recurrence, defined as a cancer recurrence in the ipsilateral breast, chest wall, or regional lymph nodes (axillary levels I-III, supraclavicular, or internal mammary)

SECONDARY OBJECTIVES FOR BOTH COHORTS

1. To compare the maximum standardized difference in arm volume between the affected arm and the unaffected arm within 24 months after completion of RNI between the two treatment arms.
2. To compare maximal acute (within 6 weeks of treatment) and late (more than 6 weeks after treatment) skin and soft tissue toxicities using the NCI CTCAE v4.0 scale between patients assigned to short versus standard RNI.
3. To compare patient-reported arm and shoulder function for the two treatment arms using the QuickDASH-9.
4. To compare patient quality of life for the two treatment arms using EQ-5D-3L and PROMIS Fatigue SF 6a.
5. To compare the peripheral blood cytokine profile at the end of radiation between patients assigned to short versus standard RNI.
6. To evaluate the effect of the peripheral blood cytokine profile at the end of radiation on developing lymphedema. (optional blood draw for a subset of patients and not applicable for the participating Cancer Network Site patients, or Orlando Health)
7. To evaluate the effect of homocysteine levels prior to radiation on developing lymphedema. (optional blood draw for a subset of patients and not applicable for the participating Cancer Network Site patients, or Orlando Health)
8. To evaluate time to distant metastasis, disease-free survival and overall survival for patients assigned to short versus standard RNI.
9. To evaluate the effect of lipid profiles prior to radiation on acute toxicity, patient reported outcomes, and the time to locoregional recurrence. (optional blood draw for a subset of patients and not applicable for the participating Cancer Network Site patients, or Orlando Health)
10. To evaluate if DNA repair capacity contributes to the presence of acute radiation related toxicity and patient-reported quality of life decrements including fatigue and arm and shoulder symptoms. (optional blood draw for a subset of patients and not applicable for the participating Cancer Network Site patients, or Orlando Health)
11. To evaluate changes in echocardiography global longitudinal strain measurements and cardiac serum biomarkers, based on measurements performed before and after RT, in patients assigned to short versus standard RNI. (optional procedure for a subset of patients and not applicable for the participating Cancer Network Site patients, or Orlando Health)
12. In a separate cohort of 50 patients who will receive RNI before surgery, to collect information on number of patients developing lymphedema within 24 months of RNI on reconstructive complications, and on patient reported quality of life, in those assigned to short versus standard RNI. Participating Cancer Network Sites, or Orlando Health, are not participating in this cohort.
13. To evaluate patient-reported financial burdens using the Economic Strain and Resilience in Cancer- Financial Well- Being instrument.
14. To determine whether radiation therapy induces de novo detectable clonal hematopoiesis mutations or alters the genetic landscape of existing clonal hematopoiesis mutations (optional blood draw for a subset of patients and not applicable for the participating Cancer Network Site patients, or Orlando Health).
15. To determine whether radiation therapy or chemotherapy among individuals with pre- and/or post-treatment clonal hematopoiesis mutations is associated with adverse treatment effects and worse oncologic outcomes (optional blood draw for a subset of patients and not applicable for the participating Cancer Network Site patients, or Orlando Health).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo hypofractionated RNI in 15 fractions 5 consecutive days a week for 3 weeks.

ARM II: Patients undergo standard RNI in 25 fractions 5 consecutive days a week for 5 weeks.

In both arms, patients undergo additional boost dose of radiation therapy in 5 or 7 fractions on consecutive days following completion of RNI.

PATIENT EVALUATION: Patients participating in the trial will have their arm measured prior to radiation, during the final week of radiation and when they return for follow up visits. Patients will be checked for any arm swelling that may develop. Patients will also fill out questionnaires before treatment and when they return for follow up visits. Patients return 3 and 6 months after radiation, then every 6 months through two and a half years after radiation and then on a yearly basis until ten and a half years after finishing radiation. At some of the follow up visits, we measure arm volume and ask participants to complete questionnaires.

ELIGIBILITY:
Inclusion Criteria, if receiving postoperative radiation therapy

* Radiation oncologist recommends radiation treatment to the supraclavicular and infraclavicular fossa (i.e. RNI).
* Pathologically-confirmed invasive breast cancer. If patients undergo upfront surgery, the pathologic stage must be T0-T3, N0-N2a or N3a. If patients receive neoadjuvant chemotherapy prior to surgery, the clinical stage must be T0-T3, N0-N2a or N3a. T4b disease is permitted if the patient undergoes breast conserving surgery.
* Treatment with mastectomy or segmental mastectomy and axillary evaluation (sentinel node evaluation, axillary sampling, or axillary lymph node dissection). If the patient has T0 disease, breast surgery is not required.
* Age 18 years or older.
* If enrolling on in the arm lymphedema assessment cohort, documentation of arm volume measurement by perometer prior to axillary surgery.
* If the patient has a history of a prior non-breast cancer, all treatment for this cancer must have been completed prior to study registration, and the patient must have no evidence of disease for this prior non-breast cancer.
* Patients must be enrolled on the trial within 24 weeks of the later of two dates: the final breast cancer surgical procedure or administration of the last cycle of cytotoxic chemotherapy. If after trial enrollment it is determined the patient requires additional cytotoxic chemotherapy or additional breast cancer surgery prior to radiation therapy the patient may stay on trial but the patient must start radiation therapy within 24 weeks of the final breast cancer surgical procedure or administration of the last cycle of cytotoxic chemotherapy.

Inclusion Criteria, if receiving preoperative radiation therapy

* Surgeon and radiation oncologist recommend preoperative radiation therapy
* Radiation oncologist recommends radiation treatment to the supraclavicular and infraclavicular fossa (i.e. RNI).
* Pathologically-confirmed invasive breast cancer. The clinical stage must be T0-T3, N0-N3b
* Planned treatment with mastectomy and axillary evaluation (sentinel node evaluation, axillary sampling, or axillary lymph node dissection).
* Planned breast reconstruction with autologous reconstruction.
* Age 18 years or older.
* If the patient has a history of a prior non-breast cancer, all treatment for this cancer must have been completed prior to study registration, and the patient must have no evidence of disease for this prior non-breast cancer.

Exclusion Criteria, if receiving postoperative radiation therapy

* Pathologic or clinical evidence for a stage T4 breast cancer. However, T4b disease is permitted if the patient undergoes breast conserving surgery.
* Pathologic or clinical evidence for a stage N2b, N3b, or N3c breast cancer (supraclavicular, or internal mammary lymph node involvement).
* Clinical or pathologic evidence for distant metastases.
* Current diagnosis of invasive breast cancer in the contralateral breast (ductal carcinoma in situ is permitted).
* Prior diagnosis of invasive breast cancer in the contralateral breast.
* If enrolling on in the arm lymphedema assessment cohort, current diagnosis of bilateral breast cancer.
* History of therapeutic irradiation to the breast, lower neck, mediastinum or other area in which there could potentially be overlap with the affected breast. Except those patients enrolled and treated on the PRECISE trial (MD Anderson 2017-0362).
* Patient is pregnant.
* Patients who are cognitively impaired. Subjects will undergo a brief physical exam including a brief exam to determine cognitive review.

Exclusion Criteria, if receiving preoperative radiation therapy

* Pathologic or clinical evidence for a stage T4 breast cancer.
* Pathologic or clinical evidence for a stage N3c breast cancer (supraclavicular lymph node involvement).
* Clinical or pathologic evidence for distant metastases.
* Current diagnosis of invasive breast cancer in the contralateral breast (ductal carcinoma in situ is permitted).
* Prior diagnosis of invasive breast cancer in the contralateral breast.
* History of therapeutic irradiation to the breast, lower neck, mediastinum or other area in which there could potentially be overlap with the affected breast. Except those patients enrolled and treated on the PRECISE trial (MD Anderson 2017-0362).
* Patient is pregnant.
* Patients who are cognitively impaired. Subjects will undergo a brief physical exam including a brief exam to determine cognitive review.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Lymphedema rate as assessed by perometry | Up to 24 months
  Will compare between patients randomized to short versus standard regional nodal irradiation (RNI). Will use a two-sided chi-squared test with a significance level of 0.05.

SECONDARY OUTCOMES:
Volume of affected and unaffected arm as assessed by perometry | Up to 126 months
  The Shapiro-Wilk test will be used to objectively assess the normality of the data and these findings will be visually confirmed by inspecting normal probability quantile-quantile plots. If the data are not normally distributed, a normalizing transformation before using t-test or a non-parametric method such as the Wilcoxon rank sum test to compare the standardized difference between the two arms at each time point may be used.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hoffman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (12):
- United States (12):
  - MD Anderson Cancer Center (Banner), Gilbert, Arizona
  - Scripps- MD Anderson Cancer, San Diego, California
  - MD Anderson Cancer Center (Banner)- Northern Colorado, Greeley, Colorado
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Community MD Anderson Cancer Center East, Indianapolis, Indiana
  - Community MD Anderson Cancer Center South, Indianapolis, Indiana
  - Community MD Anderson Cancer Center North, Indianapolis, Indiana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Ohio Health, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - UT Health San Antonio - MD Anderson Cancer Center, San Antonio, Texas

REFERENCES:
- [Derived] Schaverien MV, Singh P, Kuerer HM, Akay CL, Chavez-MacGregor M, Chu CK, Clemens MW, Qiao W, Smith BD, Hoffman KE. Comparison of Outcomes of Microsurgical Breast Reconstruction after Premastectomy and Postmastectomy Radiation Therapy. J Am Coll Surg. 2025 Oct 1;241(4):535-549. doi: 10.1097/XCS.0000000000001444. Epub 2025 Sep 16. PMID 40366003
- [Derived] Schaverien MV, Singh P, Smith BD, Qiao W, Akay CL, Bloom ES, Chavez-MacGregor M, Chu CK, Clemens MW, Colen JS, Ehlers RA, Hwang RF, Joyner MM, Largo RD, Mericli AF, Mitchell MP, Shuck JW, Tamirisa N, Tripathy D, Villa MT, Woodward WA, Zacharia R, Kuerer HM, Hoffman KE. Premastectomy Radiotherapy and Immediate Breast Reconstruction: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245217. doi: 10.1001/jamanetworkopen.2024.5217. PMID 38578640
- See also: MD Anderson Cancer Center — http://www.mdanderson.org